CLINICAL TRIAL: NCT07294729
Title: The Effects of Mulligan and Proprioceptive Neuromuscular Facilitation Techniques on Pain, Functionality, Proprioception, and Quality of Life in Individuals With Rotator Cuff Lesions
Brief Title: Mulligan and Proprioceptive Neuromuscular Facilitation Techniques in Individuals With Rotator Cuff Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Emre DANSUK, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-7892
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Syndrome; Rotator Cuff Injuries
Keywords: Rotator Cuff Syndrome; Mulligan Mobilization; Manual Therapy; Proprioceptive Neuromuscular Facilitation; Physiotherapy; Shoulder Rehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Control Groups; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group randomized controlled trial design in which participants with rotator cuff lesions are assigned to one of three groups: (1) Conventional Physiotherapy, (2) Mulligan Mobilization With Movement plus Conventional Physiotherapy, or (3) Proprioceptive Neuromuscular Facilitation plus Conventional Physiotherapy.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessors will be blinded to group allocation. The care providers administering the interventions will not be blinded due to the nature of the manual therapy techniques. Group assignments will be concealed using coded identifiers, and outcome assessments will be performed by an assessor who is unaware of the participants' treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Conventional Physiotherapy) (Active Comparator): All participants will receive a conventional physiotherapy program for 3 weeks, 4 days per week. The program includes wand exercises in all directions (10 repetitions with a 2-second end-range hold), Codman pendulum exercises in flexion, abduction, and circular motions (10 repetitions), stretching exercises held for 20 seconds for 5 repetitions in all directions, and finger-ladder exercises for flexion and abduction (10 repetitions). Strengthening exercises will be performed using elastic bands selected according to each participant's physical capacity (3 sets of 10 repetitions). All sessions will be supervised by a physiotherapist. Additionally, TENS will be applied to the painful area at 100 Hz for 20 minutes in each session.
  Interventions: Other: Control Group (Conventional Physiotherapy)
- Mulligan Group (Experimental): In the Mulligan group, the MWM (Movement With Mobilization) technique will be applied in addition to the conventional exercise program. MWM will be performed twice a week for 3 weeks in flexion, abduction, internal rotation, and external rotation. The technique will be applied before exercises. A mobilization belt will be used to provide an effective glide, and participants will first demonstrate the painful or restricted movement. The belt will be placed around the shoulder, and the joint positioned pain-free. A glide force will be applied while the participant performs the movement actively, followed by a 3-second hold at the end range. The first two sessions will include 10 repetitions; subsequent sessions will include 3 sets of 10 repetitions. Participants will be positioned supine for rotation techniques and seated for flexion and abduction.
  Interventions: Other: Control Group (Conventional Physiotherapy); Other: Mulligan Mobilization
- Proprioceptive Neuromuscular Facilitation Group (Experimental): Before the standard physiotherapy and exercise program, the "hold-relax active movement" technique will be applied to increase circulation around the joint and enhance muscle activation. This technique is based on repeated isotonic contractions that do not require continuous effort.
  The physiotherapist will first ask the participant to perform an isometric contraction in the shortened position of the agonist pattern. Then the participant will be instructed to relax, and the segment will be moved quickly and passively into the lengthened position of the antagonist pattern. The participant will then be asked to perform an isotonic contraction of the agonist pattern again.
  This sequence will be repeated several times until contraction is adequately felt in the weak muscles or until fatigue occurs. Care will be taken to ensure that the passive movement into the antagonist direction is performed smoothly and quickly.
  Interventions: Other: Control Group (Conventional Physiotherapy); Other: Proprioceptive Neuromuscular Facilitation

INTERVENTIONS:
Other: Control Group (Conventional Physiotherapy) — Participants in the control group will receive a supervised conventional physiotherapy program consisting of wand, pendulum, stretching, and finger-ladder exercises, strengthening with elastic bands, and TENS applied to the painful area at 100 Hz for 20 minutes per session.
Other: Mulligan Mobilization — Participants in the Mulligan group will receive the conventional physiotherapy program plus Mulligan Movement With Mobilization (MWM) techniques applied twice weekly before exercises. The physiotherapist will use a mobilization belt to provide joint glide while participants perform pain-free active movements in flexion, abduction, and rotation.
  Arms: Mulligan Group
Other: Proprioceptive Neuromuscular Facilitation — Participants in the PNF group will receive the conventional physiotherapy program plus PNF "hold-relax active movement" techniques applied before exercises. The physiotherapist will guide participants through repeated isometric, passive, and isotonic contractions to enhance proprioceptive input, muscle activation, and joint mobility.
  Arms: Proprioceptive Neuromuscular Facilitation Group

SUMMARY:
This study aims to compare the effects of Mulligan mobilization with movement (MWM) and Proprioceptive Neuromuscular Facilitation (PNF) techniques on pain, functionality, proprioception, and quality of life in individuals diagnosed with rotator cuff lesions. A total of 45 participants aged 30-70 years with partial supraspinatus tears confirmed by clinical and radiological assessment will be randomly assigned to three groups: conventional physiotherapy, Mulligan + conventional physiotherapy, and PNF + conventional physiotherapy. All groups will receive a standardized three-week physiotherapy program, while the Mulligan and PNF groups will additionally undergo their respective manual therapy interventions. Outcome measures will include pain intensity (VAS), shoulder range of motion, functional disability (DASH), joint position sense, and rotator cuff-specific quality of life (RC-QoL). The study seeks to determine which manual therapy approach (Mulligan or PNF) provides superior improvements in clinical outcomes compared with conventional treatment alone.

DETAILED DESCRIPTION:
Rotator cuff lesions are among the most common causes of shoulder pain and functional limitation, often resulting from overuse, degenerative changes, impaired neuromuscular control, or acute trauma. These conditions may lead to significant restrictions in daily living activities and decreased quality of life. Conservative physiotherapy remains the primary treatment approach for individuals with partial-thickness rotator cuff tears, emphasizing pain relief, range of motion restoration, neuromuscular control, and functional improvement. Recent literature suggests that manual therapy techniques, when combined with exercise programs, may enhance clinical outcomes by providing additional benefits in pain modulation, joint mobility, and sensorimotor function.

This study is designed to investigate and compare the clinical efficacy of two commonly used manual therapy techniques-Mulligan Mobilization With Movement (MWM) and Proprioceptive Neuromuscular Facilitation (PNF)-in individuals with rotator cuff lesions. Although both approaches are widely used in clinical practice, there is currently no comparative research evaluating their relative effectiveness on pain, functionality, proprioception, and quality of life. By integrating these techniques into a structured physiotherapy program, the study aims to determine whether either method provides superior therapeutic benefits.

A total of 45 participants aged 30-70 years with a confirmed diagnosis of partial supraspinatus tear will be included. Diagnosis will be established by a physical medicine and rehabilitation specialist and verified through appropriate imaging techniques. Participants will be randomly allocated into three groups: (1) Conventional Physiotherapy (Control), (2) Mulligan + Conventional Physiotherapy, and (3) PNF + Conventional Physiotherapy. All groups will receive a standardized physiotherapy program consisting of wand exercises, Codman pendulum exercises, stretching, finger-ladder exercises, strengthening with elastic bands tailored to individual capability, and TENS applied at 100 Hz for 20 minutes per session. This program will be administered four times per week for three weeks under physiotherapist supervision.

In the Mulligan group, the MWM technique will be applied prior to the exercise program. The intervention will target shoulder flexion, abduction, internal rotation, and external rotation. Using a mobilization belt to optimize joint gliding, the therapist will guide the participant through active, pain-free movements while applying a sustained accessory glide. The technique will initially be performed for 10 repetitions in the first two sessions and progressed to 3 sets of 10 repetitions in later sessions.

In the PNF group, a "hold-relax active movement" approach will be used to enhance proprioceptive input, neuromuscular activation, and functional movement patterns. Participants will perform isometric contractions in the shortened range of the agonist muscle, followed by relaxation and quick passive movement into the elongated range of the antagonist pattern. They will then perform isotonic contractions of the agonist. This cycle will be repeated several times until adequate muscle activation or fatigue is achieved. PNF will also be performed prior to the conventional exercise program.

Outcome measurements will be performed at baseline and at the end of the three-week intervention period. Pain intensity will be assessed using the Visual Analog Scale (VAS), and shoulder joint range of motion will be measured using the Goniometer Pro smartphone application, which has demonstrated good validity and reliability. Functional disability will be evaluated using the Turkish version of the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire, while proprioception will be measured through joint position sense testing at 60 degrees of flexion and abduction using Goniometer Pro. Quality of life will be assessed through the Rotator Cuff Quality of Life (RC-QoL) questionnaire, which has been validated for Turkish-speaking patients with rotator cuff pathology.

Statistical analyses will be conducted using SPSS 25.0. Normality will be tested through skewness-kurtosis values. Depending on distribution, within-group comparisons will utilize paired t-tests or Wilcoxon signed-rank tests; between-group comparisons will use one-way ANOVA or Kruskal-Wallis tests. When significant group differences are identified, appropriate post-hoc analyses will be performed. A significance level of p < 0.05 will be adopted.

This study is expected to contribute important evidence regarding the comparative effectiveness of Mulligan MWM and PNF techniques for rotator cuff lesions. The findings may support clinicians in selecting the most beneficial manual therapy approach to optimize patient outcomes in terms of pain reduction, functional capacity, proprioceptive accuracy, and overall quality of life. The results may also guide future research focusing on combined manual therapy and exercise interventions for shoulder pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between 30 and 70 years of age.
* A diagnosis of partial supraspinatus tear made by a physical medicine and rehabilitation s-specialist.
* Confirmation of the diagnosis through radiological imaging methods.
* No history of any shoulder surgery.
* Shoulder symptoms persisting for more than 4 weeks.

Exclusion Criteria:

* Individuals who are unable to cooperate or who have mental health problems.
* Individuals who have participated in any shoulder-related physiotherapy program within the last 3 months.
* Individuals with other musculoskeletal conditions that may affect the shoulder region.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Joint Position Sense | 3 weeks
  Joint position sense will be assessed using the Becure Extremity ROM system. Joint position sense will be assessed at 60 degrees of shoulder flexion and shoulder abduction. While standing, the participant will first be asked to lift the arm with eyes open and memorize the position at 60 degrees. Then, with eyes closed, the participant will be instructed to raise the arm to the same position reached when the eyes were open. The shoulder angle obtained with eyes closed will be recorded. The difference between the angles measured with eyes open and eyes closed will be considered the joint position sense error. This method will be performed at 60 degrees of both flexion and abduction.

SECONDARY OUTCOMES:
Pain (VAS Score) | 3 weeks
  The Visual Analog Scale (VAS) is a commonly used method for assessing pain intensity. Participants will be asked to mark the level of pain they feel on a 100-mm line. The lower end of the line represents low pain intensity, while the upper end indicates high pain intensity.
Range of Motion (Shoulder Flexion, Abduction, Internal and External Rotation Measured in Degrees) | 3 weeks
  The shoulder range of motion of the participants will be measured using the Goniometer Pro smartphone application. Flexion and abduction will be assessed within a range of 0-180 degrees, and internal and external rotation within a range of 0-90 degrees.
Disability (DASH Questionnaire Score) | 3 weeks
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is used to assess physical disability and functional status in upper extremity injuries. The questionnaire consists of three subcategories. The first section contains 30 items evaluating the patient's functional status and symptoms. Of these 30 items, 21 assess daily living activities, 5 assess symptoms (pain, pain with activity, tingling, weakness, and movement limitations), and the remaining 4 assess social function, work, sleep, and self-confidence. The work module consists of 4 additional items evaluating the individual's work-related function. Each question is scored using a 5-point Likert scale (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: severe difficulty, 5: unable to do). Higher scores indicate greater disability.
Quality of Life (RC-QoL Score) | 3 weeks
  The Rotator Cuff Quality of Life (RC-QoL) questionnaire is a condition-specific assessment tool designed to measure quality of life in individuals with rotator cuff pathology. The scale consists of 34 items organized into five domains: physical symptoms, work-related activities, activities of daily living, social functioning, and emotional well-being. Each question is scored on a scale from 0 to 100, where "0" indicates severe pain and "100" indicates no pain. Higher scores reflect better quality of life. The total score is calculated by summing the item scores, dividing by the number of answered items, and expressing the result as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Dansuk, PhD, Principal Investigator — Medipol University
Locations (1):
- Emre Dansuk, Istanbul, Beykoz, Turkey (Türkiye)